CLINICAL TRIAL: NCT06365892
Title: Effectiveness of Conditioning + Open-label Placebo for the Management of Pain in Children Who Undergo Surgical Treatment of Idiopathic Scoliosis
Brief Title: Open-label Placebo (COLP) for Pain in Adolescent Idiopathic Scoliosis (AIS) Surgery+Surgical Treatment of Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-36548
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Conditioning with Open-Label Placebo (COLP)
MeSH Terms: interventions — Sugars; Therapeutics

STUDY DESIGN:
Intervention Model Description: Both arms - Open-label Placebo (COLP) and Treatment As Usual (TAU)
Masking Description: Blinding of patients and providers will not be feasible due to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open-label Placebo (COLP) (Experimental): Placebo will be supplied as a 330mg tablet (manufactured by Consolidated Midland Corporation). Each oral opioid dose is a 5mg Oxycodone tablet. Patients will take placebo with each oral opioid intake and 3 additional times per day beginning on POD 1. Investigator shall never prescribe ibuprofen. Investigator shall always prescribe Tylenol 625mg every 8hrs (PRN).
  Interventions: Other: open-label placebo; Other: Treatment as usual
- Treatment As Usual (TAU) (Experimental): Treatment As Usual (TAU) subjects will receive equal access to opioid and non-opioid analgesics. The preferred oral opioid dose is a 5mg Oxycodone pill. Subjects will take a placebo with each oral opioid dose and additional three times per day beginning on POD 1.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: open-label placebo — Placebo will be supplied as a 330mg tablet (manufactured by Consolidated Midland Corporation). Patients will take placebo with each oral opioid intake and 3 additional times per day beginning on POD 1.
  Other Names: Inactive drug, Inactive medicine, Inactive substance, Sugar Pill Test Substance
  Arms: Open-label Placebo (COLP)
Other: Treatment as usual — Each oral opioid dose is a 5mg Oxycodone tablet. Investigator shall never prescribe ibuprofen. Investigator shall always prescribe Tylenol 625mg every 8hrs (PRN).

SUMMARY:
This study aims to investigate the effects of conditioning with open-label placebos on standard postoperative treatment for patients undergoing surgery for idiopathic scoliosis in a randomized controlled, 6-week trial with 64 AIS patients randomly assigned to one of two arms: Open-label Placebo (COLP) + treatment as usual TAU / TAU control. The study involves collecting data from your child's medical record. At each regular clinic visit, the patient clinical data will be collected by the research coordinator. Surveys will be collected including:• PROMIS for the age group 10 to 18 years.

DETAILED DESCRIPTION:
Interventional (clinical trial): Subject will be randomly assigned using permuted blocks (block size of 4). Before usage, random assignments will be created, stored in sealed envelopes, and numbered (1, 2, etc.). There will be stratified randomization: Later on, stratification will be incorporated into the analysis. 32 people will be in the group taking the placebo pills in addition to standardized treatment and 32 people will be in the group with standardized treatment alone.

Hypothesis: Open-label Placebo (COLP) < treatment as usual (TAU) control. Secondary Aims Analysis Plan: There are three secondary aims in this study.

Aim 1. To determine whether 6 weeks of Open-label Placebo (COLP) results in significantly reduced opioid consumption compared to treatment as usual. To test this aim, the investigators will conduct a t-test comparing mean opioid use over the 6 weeks of follow up. In secondary analyses, the investigators will adjust for any baseline factors including gender, age, symptom severity or type of surgery that could be a confounding variable.

1a. To determine if 6 weeks of Open-label Placebo (COLP) results in reduced opioid consumption compared to treatment as usual. Hypothesis: Open-label Placebo (COLP) < treatment as usual (TAU) control.

Secondary Aims Analysis Plan: There are three secondary aims in this study.

Secondary Aim 1: Determine if there are significant differences in time to independence with physical therapy, length of stay, time to return to school, urinary retention, constipation, oxygen requirement, and number of contacts with medical team in Open-label Placebo (COLP) compared to treatment as usual (TAU).

Secondary Aim 2: Determine if there is an association between preoperative pain catastrophization, kinesiophobia, positive/negative affect, anxiety, and/or depression and response to Open-label Placebo (COLP) and/or treatment as usual (TAU).

Secondary Aim 3: Determine if there is an association between postoperative PROMIS scores, anxiety, and/or depression in open-label placebo (COLP) compared to treatment as usual (TAU).

Primary Objectives The primary objectives of this study are to: (1) to determine whether 6 weeks of conditioning with open-label placebo (COLP) results in reduced opioid consumption (amount and duration) compared to treatment as usual (TAU) control and (2) to determine whether 6 weeks of Open-label Placebo (COLP) compared to treatment as usual (TAU) results in different clinical outcomes.

Secondary Objectives

* To determine whether open-label placebo (COLP) affects anxiety and/or depression.
* To determine whether open-label placebo (COLP) affects length of stay, opioid side effects, time to independence with physical therapy, and/or number of contacts with medical team.
* To determine if there is an association between pain catastrophizing, kinesiophobia, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, patients must meet all of the following inclusion criteria:

1. Diagnosis of idiopathic spine deformity.
2. Age >10 and <18 years.
3. Primary procedure.
4. Guardian provides signed and dated informed consent and understand the nature of the study sufficiently to allow completion of all study assessments.
5. Patient provides assent.
6. Fusion and fusionless instrumented spine surgery.

Exclusion Criteria:

If any of the following exclusion criteria are met, the patient is not eligible for the study:

1. Non-idiopathic scoliosis, such as neuromuscular or syndrome.
2. Revision procedure.
3. Self-reported pregnancy or planned pregnancy within the next two months.
4. Have a history of drug, excluding nicotine or caffeine, or alcohol abuse within 2 years of entry into the study
5. Already taking opioids.
6. Abnormal physical examination.
7. Inability to speak or read English
8. Patient declines participation.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The total amount of opioids consumed in oral morphine equivalents (OMEs) following surgery | from admission to 6 weeks post-operatively
  Oral morphine equivalents (OMEs) are values that represent the potency of an opioid dose relative to morphine. Using OMEs provides a standardized method for converting between various opiate medications. Each oral opioid dose is a 5mg Oxycodone tablet prescribed 6 times per day pro re nata. Participants will record the number of oral opioids taken each day for 6 weeks following surgery beginning on Post-op Day 1 (POD1). This data will be collected and converted into OMEs for comparison.

SECONDARY OUTCOMES:
Weekly level of mobility and change from baseline in mobility on the Patient-Reported Outcome Measurement Information System (PROMIS) Numeric Rating Scale Pediatric Mobility Short Form 7a at week 6. | weekly from admission to 6 weeks post-operatively
  the PROMIS Pediatric Mobility SF 7a is a validated, self-reported instrument that consists of 7 items rating mobility on average over the past 7 days from 4 (With no trouble) to 0 (not able to do). Weekly level of mobility = mobility score reported at each week Change = (Week 6 Score - Baseline Score).
Weekly level of anxiety and change from baseline in anxiety levels on the Patient-Reported Outcome Measurement Information System (PROMIS) Numeric Rating Scale Anxiety Short Form 8a at week 6. | weekly from admission to 6 weeks post-operatively
  the PROMIS Anxiety SF 8a is a validated, self-reported instrument that consists of 8 items rating anxiety on average over the past 7 days from 1 (never) to 5 (almost always). Weekly level of anxiety = anxiety score reported at each week Change = (Week 6 Score - Baseline Score).
Weekly level of depressive symptoms and change from baseline in depressive symptoms on the Patient-Reported Outcome Measurement Information System (PROMIS) Numeric Rating Scale Depressive Symptoms Short Form 8a at week 6. | weekly from admission to 6 weeks post-operatively
  the PROMIS Depressive Symptoms SF 8a is a validated, self-reported instrument that consists of 8 items rating depressive symptoms on average over the past 7 days from 1 (never) to 5 (almost always).
  Weekly level of depressive symptoms = depressive symptoms score reported at each week Change = (Week 6 Score - Baseline Score).
The duration of time in days following surgery until patients establish Independence with Physical Therapy | from admission to final physical therapy assessment, up to 6 weeks
  Participants will be treated by physical therapy services after surgery until their physical therapist determines that they no longer require physical therapy services. Duration of time to independence with physical therapy is equal to the POD # where physical therapist determines formal PT is no longer required.
The length of time in days following surgery until discharge from the hospital | from admission to discharge, up to 6 weeks
  Participants will be admitted to the hospital following surgery until they are cleared for discharge from a medical standpoint.
  Length of stay = POD # that patient is discharged
The length of time in days following surgery until participant returns to school | from admission to date of return to school, up to 6 weeks post-operatively
  Participants will record the date on which they return to school after surgery. The POD # on date of return to school = the length of time to return to school. The amount of time it takes to return to school can be used as a proxy for whether participants are struggling with their pain or not.
Whether participants experience urinary retention following surgery. | during hospitalization until discharge, up to 6 weeks
  Participants will be assessed in hospital to determine whether or not they experience urinary retention post-surgery, a potential side effect of opioid consumption. The urinary retention determination will be a yes/no answer.
Whether participants experience constipation measured by the number of days between surgery and first bowel movement | from admission to date of first bowel movement, up to 6 weeks post-operatively
  Participants will record the number of days between surgery and first bowel movement to assess whether they experience constipation, a potential side effect of opioid consumption.
Whether participants experience an oxygen requirement and the duration of the requirement following surgery. | during hospitalization until discharge, up to 6 weeks
  Participants will be assessed in hospital for whether or not they have an oxygen requirement and the duration of requirement. The oxygen requirement will be a yes/no answer. If yes, the number of days that oxygen is required will be recorded for the duration.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Diab, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho C, Caetano JM, Cunha L, Rebouta P, Kaptchuk TJ, Kirsch I. Open-label placebo treatment in chronic low back pain: a randomized controlled trial. Pain. 2016 Dec;157(12):2766-2772. doi: 10.1097/j.pain.0000000000000700. PMID 27755279
- [Background] Blease C, Colloca L, Kaptchuk TJ. Are open-Label Placebos Ethical? Informed Consent and Ethical Equivocations. Bioethics. 2016 Jul;30(6):407-14. doi: 10.1111/bioe.12245. Epub 2016 Feb 3. PMID 26840547
- [Background] von Wernsdorff M, Loef M, Tuschen-Caffier B, Schmidt S. Effects of open-label placebos in clinical trials: a systematic review and meta-analysis. Sci Rep. 2021 Feb 16;11(1):3855. doi: 10.1038/s41598-021-83148-6. PMID 33594150
- [Background] Kirchhof J, Petrakova L, Brinkhoff A, Benson S, Schmidt J, Unteroberdorster M, Wilde B, Kaptchuk TJ, Witzke O, Schedlowski M. Learned immunosuppressive placebo responses in renal transplant patients. Proc Natl Acad Sci U S A. 2018 Apr 17;115(16):4223-4227. doi: 10.1073/pnas.1720548115. Epub 2018 Apr 2. PMID 29610294
- [Background] Ader R, Mercurio MG, Walton J, James D, Davis M, Ojha V, Kimball AB, Fiorentino D. Conditioned pharmacotherapeutic effects: a preliminary study. Psychosom Med. 2010 Feb;72(2):192-7. doi: 10.1097/PSY.0b013e3181cbd38b. Epub 2009 Dec 22. PMID 20028830
- [Background] Doering BK, Rief W. Utilizing placebo mechanisms for dose reduction in pharmacotherapy. Trends Pharmacol Sci. 2012 Mar;33(3):165-72. doi: 10.1016/j.tips.2011.12.001. Epub 2012 Jan 25. PMID 22284159
- [Background] Sandler AD, Glesne CE, Bodfish JW. Conditioned placebo dose reduction: a new treatment in attention-deficit hyperactivity disorder? J Dev Behav Pediatr. 2010 Jun;31(5):369-75. doi: 10.1097/DBP.0b013e3181e121ed. PMID 20495473
- [Background] Nurko S, Saps M, Kossowsky J, Zion SR, Di Lorenzo C, Vaz K, Hawthorne K, Wu R, Ciciora S, Rosen JM, Kaptchuk TJ, Kelley JM. Effect of Open-label Placebo on Children and Adolescents With Functional Abdominal Pain or Irritable Bowel Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):349-356. doi: 10.1001/jamapediatrics.2021.5750. PMID 35099543
- [Background] Flowers KM, Patton ME, Hruschak VJ, Fields KG, Schwartz E, Zeballos J, Kang JD, Edwards RR, Kaptchuk TJ, Schreiber KL. Conditioned open-label placebo for opioid reduction after spine surgery: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1828-1839. doi: 10.1097/j.pain.0000000000002185. PMID 33449503
- [Derived] Furie KS, James K, Kaptchuk TJ, Diab M. Effectiveness of conditioning + open-label placebo for post-operative pain management in adolescent idiopathic scoliosis. Pain Manag. 2025 Jul;15(7):363-371. doi: 10.1080/17581869.2025.2520148. Epub 2025 Jun 19. PMID 40536435
- See also: Mohammad Diab, MD — https://profiles.ucsf.edu/mohammad.diab